CLINICAL TRIAL: NCT02989337
Title: Endothelial Dysfunction in Hyperemesis Gravidarum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erdem Sahin, Principal Investigator, Kayseri Education and Research Hospital
Other Study IDs: 2016/579
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Hyperemesis; Gravidarum, With Dehydration
Keywords: Hyperemesis Gravidarum; Inflammatory adhesion molecules; Dehydration
MeSH Terms: conditions — Hyperemesis Gravidarum; Dehydration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- hyperemesis gravidarum with dehydration: The first group was formed of the patients diagnosed hyperemesis gravidarum with dehydration
- Control group: The control group was formed of the patients who were healthy pregnant women admitted to the clinic just for routine examination without any symptoms

SUMMARY:
The purpose of the study is to determine serum inflammatory adhesion molecules levels in hyperemesis gravidarum

DETAILED DESCRIPTION:
The study population consisted of 2 groups; (1) the hyperemesis gravidarum group, consist of 25 pregnant women who developed dehydration due to HG between 6 and 13 gestational weeks and between 18 and 35 years (2) the normal pregnancy group, consisting of 25 pregnant women.

HG was defined according to the fallowing American College of Obstetricians and Gynecologists (ACOG) criteria; severe nausea and vomiting resulted in 5% weight loss with regard to pre-gestation or vomiting more than 3 times and 3-5 % weight loss with ketonuria. The diagnosis of dehydration was clinically defined and patients with moderate and severe dehydration were included in the study. As clinical findings; Weight loss, capillary recall time, dry mucous membranes, dry eye, pulse rate, systolic blood pressure, respiration, skin turgor deterioration and urine output were evaluated.

Other pathologies causing nausea and vomiting like; gastroenteritis, gastroparesis, gall duct diseases, hepatitis, peptic ulcers, appendicitis, pyelonephritis, ovarian torsion, urinary tract stones, diabetic ketoacidosis, hyperthyroidism, hyperparathyroidism, migraine, pseudo tumor cerebra, vestibular diseases were excluded from the study.Patients were excluded from the study in the presence of pregestational diabetes chronic hypertension, chronic liver and renal failure, preeclampsia history, multiple pregnancy, hyperlipidemia, hypercholesterolemia, obesity, tobacco use, NSAID drug use, infection within the last three months and surgery within the last month that could cause endothelial dysfunction.

Blood and urine specimens were collected from the patients with HG during hospitalization and during regular clinic visits in control group. The 2mL of blood samples were withdrawn into serum-separating tubes for the measurements of serum biochemical parameters and 2 mL blood samples were withdrawn into EDTA containing tubes for measurement serum hemoglobin and hematocrit levels. Early-morning urine samples were collected from study population. These blood and urine samples were analyzed in same day for Kayseri Education and Research hospital biochemical clinics. In addition 2mL of blood samples were withdrawn into serum-separating tubes for analyzing serum sVEGFR-1, sVCAM-1, sE-selectin and sICAM-1 levels. All of the serum were stored at -80°C in nonadsorbable tubes. After three months for stored first blood sample, serum sVEGFR-1, sVCAM-1, sE-selectin and sICAM-1 levels were determined by an enzyme linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* 6-13 gestational weeks
* between 18-35 years of age
* Single pregnancy
* Dehydration due to HG

Exclusion Criteria:

Other pathologies causing nausea and vomiting;

* gastroenteritis
* gastroparesis
* gall duct diseases
* hepatitis
* peptic ulcers
* appendicitis
* pyelonephritis
* urinary tract stones
* hyperthyroidism
* hyperparathyroidism
* migraine
* vestibular diseases

Patients were excluded from the study in the presence of parameters that may cause endothelial dysfunction such as;

* pregestational diabetes
* chronic hypertension
* chronic liver and renal failure
* preeclampsia history
* multiple pregnancy
* hyperlipidemia
* hypercholesterolemia
* obesity
* tobacco use
* NSAID drug use
* infection within the last three months
* surgery within the last month

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of 2 groups; (1) the hyperemesis gravidarum group, consist of 25 pregnant women who developed dehydration due to HG between 6 and 13 gestational weeks and between 18 and 35 years (2) the normal pregnancy group, consisting of 25 pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Serum inflammatory adhesion molecules in hyperemesis gravidarum | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Erdem SAHİN, Principal Investigator — Kayseri Training and Research Hospital
Locations (1):
- Kayseri Training and Research Hospital, Kayseri, Turkey (Türkiye)